CLINICAL TRIAL: NCT00234494
Title: A Phase II Trial of Cisplatin, Gemcitabine and Bevacizumab in Combination for Metastatic Transitional Cell Cancer: Hoosier Oncology Group GU04-75
Brief Title: Cisplatin, Gemcitabine and Bevacizumab in Combination for Metastatic Transitional Cell Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Christopher Sweeney, MBBS (Other)
Collaborators: Genentech, Inc. (Industry); Eli Lilly and Company (Industry); Walther Cancer Institute (Other); Hoosier Cancer Research Network (Other)
Responsible Party: Sponsor-Investigator, Christopher Sweeney, MBBS, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOG GU04-75
Record Dates: First submitted 2005-10-05; First posted 2005-10-07 (Estimated); Results first posted 2016-03-14 (Estimated); Last update posted 2016-03-14 (Estimated); Status verified 2016-02

CONDITIONS: Bladder Cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Cisplatin; Gemcitabine; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Group Assignment (Experimental): Cisplatin + Gemcitabine + Bevacizumab
  Interventions: Drug: Cisplatin; Drug: Gemcitabine; Drug: Bevacizumab

INTERVENTIONS:
Drug: Cisplatin — Cisplatin 70 mg/m2, day 1
Drug: Gemcitabine — Gemcitabine 1250 mg/m2, day 1 and 8
Drug: Bevacizumab — Bevacizumab 15mg/kg, day 1

SUMMARY:
Cisplatin is a very important agent for the treatment of TCC as it has a single agent response rate of approximately 15%. However, it has been most important as a part of combination chemotherapy, MVAC initially and now in combination with gemcitabine. Single agent gemcitabine has demonstrated an overall response rate (ORR) of approximately 25%, including some complete responses (CR), with minimal toxicity in patients with advanced bladder cancer. Bevacizumab, a murine anti-human VEGF monoclonal antibody, has been advanced for use in combination with cytotoxic chemotherapy to delay time to disease progression in patients with metastatic solid tumors.

This trial is designed to further assess the efficacy, safety and tolerability of this regimen in this patient population.

DETAILED DESCRIPTION:
OUTLINE: This is a multi-center study.

* Cisplatin 70 mg/m2 Day 1
* Gemcitabine 1250 mg/m2 Day 1 and 8
* Bevacizumab 15 mg/kg Day 1

Review toxicity every cycle (every 3 weeks) Review for radiographic response every 2 cycles (every six weeks)

Progressive disease = off protocol therapy

Patients will be treated for up to a maximum of 8 cycles of cisplatin and gemcitabine (24 weeks of therapy). If a patient has not progressed by the end of 24 weeks (completion of cisplatin and gemcitabine), then patient will be treated with bevacizumab at 15 mg/kg every three weeks for a maximum of 12 months of bevacizumab therapy (since study entry).

If at any time patient has undue toxicity or progressive disease, patient will be removed from the study and followed until progression and for survival.

If the patient has Grade 3 or 4 neurotoxicity and/or the creatinine rises above 2.0, then the cisplatin will be discontinued and the patient continued on study and treated with gemcitabine and bevacizumab at the same dose and schedule.

ECOG Performance Status 0 or 1

Hematopoietic:

* White blood cell count > 3000/mm3
* Absolute neutrophil count (ANC) > 1500 mm/3
* Platelet count > 100,000/mm3
* Hemoglobin > 8 g/dL (may be transfused or receive erythropoietin support to maintain or exceed this level).
* INR < 1.5
* No full dose/therapeutic anticoagulation with either low molecular weight heparin or unfractionated heparin or coumadin

Hepatic:

* Total bilirubin of <1.5 mg/dL
* ALT <5 times upper limit of normal for subjects with documented liver metastases; <2.5 times the upper limit of normal for subjects without evidence of liver metastases.

Renal:

* Serum creatinine of < 1.5 mg/dL.
* Urine protein:creatinine ratio < 1.0 at screening

Cardiovascular:

* No history of myocardial infarction or stroke within the last 6 months
* No uncontrolled hypertension (blood pressure of >160 systolic and/or 110 diastolic mmHg on medication)
* No unstable angina, New York Heart Association (NYHA) Grade II or greater congestive heart failure
* No unstable symptomatic arrhythmia requiring medication (subjects with chronic atrial arrhythmia, i.e., atrial fibrillation or paroxysmal supraventricular tachycardia are eligible), or clinically significant peripheral vascular disease.

Pulmonary:

* Not specified

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated or relapsed locally advanced or metastatic transitional cell carcinoma of the bladder. (Patients with pathology showing ANY component of non-transitional cell histology are not eligible).
* Relapsed patients may have received prior chemotherapy ≥ one year prior to study registration as part of a neoadjuvant or adjuvant regimen and must not have had intervening therapy from the end of that treatment until study entry.
* Measurable disease as per RECIST.
* Prior radiation therapy, immunotherapy, cytokine, biologic or vaccine therapy must be greater than 28 days prior to being registered for protocol therapy,

Exclusion Criteria:

* No known central nervous system metastasis. (imaging of brain only required if clinically indicated)
* No prior organ allograft.
* No history of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications.
* No evidence of bleeding diathesis or coagulopathy.
* No history of serious, non-healing wound, ulcer or bone fracture
* No history of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to being registered for protocol therapy.
* No prior history of malignancy in the past 5 years with the exception of basal cell and squamous cell carcinoma of the skin. Other cancers with low potential for metastasis, such as in situ cancers (e.g., Grade 1, TA TCC (low grade superficial bladder cancer), colonic polyp with focus of adenocarcinoma) can also be enrolled after approval from the study chair.
* No major surgical procedure, open biopsy, or significant traumatic injury less than 28 days prior to being registered for protocol therapy.
* Patients are not eligible if the need for any major surgical procedure is anticipated during the course of the study.
* Any minor surgical procedures, fine needle aspirations or core biopsies must be greater than 7 days prior to being registered for protocol therapy except procedures to secure a vascular access device which must be greater than 7 days prior to the start of protocol therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2005-11; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Sweeney, M.B.B.S., Study Chair — Hoosier Oncology Group, LLC
Locations (11):
- United States (11):
  - University of Chicago, Chicago, Illinois
  - Medical & Surgical Specialists, LLC, Galesburg, Illinois
  - Oncology Hematology Associates of SW Indiana, Evansville, Indiana
  - Fort Wayne Oncology & Hematology, Inc, Fort Wayne, Indiana
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Quality Cancer Center (MCGOP), Indianapolis, Indiana
  - Arnett Cancer Care, Lafayette, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - AP&S Clinic, Terre Haute, Indiana
  - Siteman Cancer Center, St Louis, Missouri
  - Oncology Hematology Care, Inc., Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hahn NM, Stadler WM, Zon RT, Waterhouse D, Picus J, Nattam S, Johnson CS, Perkins SM, Waddell MJ, Sweeney CJ; Hoosier Oncology Group. Phase II trial of cisplatin, gemcitabine, and bevacizumab as first-line therapy for metastatic urothelial carcinoma: Hoosier Oncology Group GU 04-75. J Clin Oncol. 2011 Apr 20;29(12):1525-30. doi: 10.1200/JCO.2010.31.6067. Epub 2011 Mar 21. PMID 21422406
- See also: Hoosier Cancer Research Network Homepage — http://www.hoosiercancer.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Group Assignment
Started | 45
Completed | 43
Not Completed | 2
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Arm/Group | Single Group Assignment
Number analyzed (Participants) | 43
Age, Customized [Median (Full Range); unit: years]
  Age | 66 [41 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 33
Region of Enrollment [Number; unit: participants]
  United States | 43
Body Mass Index, kg/m2 [Median (Full Range); unit: kg/m2] | 27.7 [19.1 to 44]
Creatinine, mg/dL [Median (Full Range); unit: mg/dL] | 1.1 [0.6 to 1.4]
WBC Count [Median (Full Range); unit: K/ul] | 7600 [4100 to 22000]
Hemoglobin [Median (Full Range); unit: g/dL] | 13.0 [9.1 to 15.6]
Platelet count [Median (Full Range); unit: platelets per ul] | 291000 [139000 to 770000]
Number of metastatic sites [Median (Full Range); unit: number of metastatic sites] | 2 [0 to 6]
Prior cystectomy [Number; unit: participants]
  Yes | 17
  No | 26
Eastern Cooperative Oncology Group (ECOG) Performance Status [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) from 0-5 that describes a patient's level of functioning where 0=Fully active, able to carry on all pre-disease performance without restriction and 5=Dead:
  participants
    ECOG 0 | 26
    ECOG 1 | 17
Metastatic Site Locations [Number; unit: number of metastatic sites per location]
  Any lymph node | 39
  Pelvic/abdominal lymph node | 27
  Any visceral metastases | 30
  Lung | 18
  Bone | 11
Modified Bajorin risk group [Number; unit: participants] — Modified Bajorin risk groups were defined as follows:PS0 and no visceral metastases(lowrisk); PS1 and no visceral metastases or PS 0 and visceral metastases (intermediate risk); and PS
  1 and visceral metastases (high risk)
  participants
    Good risk | 8
    Intermediate risk | 23
    Poor risk | 12

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: - To determine the progression free survival of patients with metastatic transitional cell cancer treated with cisplatin, gemcitabine and bevacizumab.
Time Frame: 36 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Single Group Assignment
Number analyzed (Participants) | 43
months | 8.2 [6.8 to 10.3]

2. Secondary Outcome: Overall Survival Time
Description: To estimate overall survival time in months.
Time Frame: 36 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Single Group Assignment
Number analyzed (Participants) | 43
months | 19.1 [12.4 to 22.7]

3. Secondary Outcome: Estimate Response Rates
Description: To estimate rate of partial response (PR), complete response (CR) and overall response (PR plus CR).
Time Frame: 36 months
Measure: Number; unit: percentage of participants
Arm/Group | Single Group Assignment
Number analyzed (Participants) | 43
percentage of participants
  complete reponse | 19
  partial reponse | 53
  overall response | 72

4. Secondary Outcome: Duration of Response for Responding Patients
Description: To estimate duration of response for responding patients.
Time Frame: 36 months
Population: Data for this secondary outcome measure was not collected or analyzed.
Arm/Group | Single Group Assignment
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Single Group Assignment
Serious Adverse Events (participants affected / at risk) | 26/45
Other Adverse Events (participants affected / at risk) | 43/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Group Assignment (N=45)
CARDIAC GENERAL - OTHER (SPECIFY, __) (Cardiac disorders) | 2 (2)
CONFUSION (Nervous system disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 2 (2)
DEHYDRATION (Gastrointestinal disorders) | 1 (1)
FEBRILE NEUTROPENIA (ANC <1.0 X 10E9/L, FEVER >=38.5 DEGREES C) (Infections and infestations) | 1 (1)
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 1 (3)
HEMOGLOBIN (Blood and lymphatic system disorders) | 1 (1)
HEMORRHAGE, CNS (Nervous system disorders) | 2 (2)
HEMORRHAGE, GI / ABDOMEN NOS (Gastrointestinal disorders) | 1 (1)
INFECTION WITH GRADE 3 OR 4 NEUTROPHILS (ANC <1.0 X 10E9/L) / URINARY TRACT NOS (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / CATHETER-RELATED (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / SCROTUM (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / URINARY TRACT NOS (Infections and infestations) | 3 (3)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / EXTRAOCULAR (Eye disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (1)
OBSTRUCTION, GU / URETER (Renal and urinary disorders) | 1 (1)
PAIN / ABDOMEN NOS (Gastrointestinal disorders) | 1 (1)
PAIN / BACK (General disorders) | 1 (1)
PHLEBITIS (INCLUDING SUPERFICIAL THROMBOSIS) (Vascular disorders) | 1 (1)
PLATELETS (Blood and lymphatic system disorders) | 1 (1)
PROTEINURIA (Investigations) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 2 (2)
SEIZURE (Nervous system disorders) | 1 (1)
SUPRAVENTRICULAR AND NODAL ARRHYTHMIA / SINUS BRADYCARDIA (Cardiac disorders) | 1 (1)
THROMBOSIS/THROMBUS/EMBOLISM (Vascular disorders) | 5 (6)
VESSEL INJURY-ARTERY / AORTA (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Group Assignment (N=45)
ALBUMIN, SERUM-LOW (HYPOALBUMINEMIA) (Investigations) | 1 (1)
ALKALINE PHOSPHATASE (Investigations) | 1 (1)
ALLERGIC RHINITIS (INCLUDING SNEEZING, NASAL STUFFINESS, POSTNASAL DRIP) (Immune system disorders) | 2 (6)
ALT, SGPT (SERUM GLUTAMIC PYRUVIC TRANSAMINASE) (Investigations) | 1 (1)
ANOREXIA (Gastrointestinal disorders) | 26 (38)
ARTHRITIS (NON-SEPTIC) (Musculoskeletal and connective tissue disorders) | 2 (2)
AST, SGOT(SERUM GLUTAMIC OXALOACETIC TRANSAMINASE) (Investigations) | 1 (1)
AUDITORY/EAR - OTHER (SPECIFY, __) (Ear and labyrinth disorders) | 1 (1)
BLOOD/BONE MARROW - OTHER (SPECIFY, __) (Blood and lymphatic system disorders) | 2 (3)
CALCIUM, SERUM-HIGH (HYPERCALCEMIA) (Investigations) | 2 (2)
CALCIUM, SERUM-LOW (HYPOCALCEMIA) (Investigations) | 1 (2)
CARDIAC GENERAL - OTHER (SPECIFY, __) (Cardiac disorders) | 1 (1)
CATARACT (Eye disorders) | 1 (1)
CHOLESTEROL, SERUM-HIGH (HYPERCHOLESTREMIA) (Investigations) | 1 (1)
CONFUSION (Nervous system disorders) | 2 (2)
CONSTIPATION (Gastrointestinal disorders) | 25 (32)
CONSTITUTIONAL SYMPTOMS - OTHER (SPECIFY, __) (General disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 10 (15)
CREATININE (Investigations) | 12 (17)
DEHYDRATION (Gastrointestinal disorders) | 2 (3)
DERMATOLOGY/SKIN - OTHER (SPECIFY, __) (Skin and subcutaneous tissue disorders) | 3 (3)
DIARRHEA (Gastrointestinal disorders) | 13 (17)
DISTENSION/BLOATING, ABDOMINAL (Gastrointestinal disorders) | 1 (1)
DIZZINESS (Nervous system disorders) | 4 (4)
DRY MOUTH/SALIVARY GLAND (XEROSTOMIA) (Gastrointestinal disorders) | 1 (1)
DYSPNEA (SHORTNESS OF BREATH) (Respiratory, thoracic and mediastinal disorders) | 12 (20)
EDEMA: LIMB (Blood and lymphatic system disorders) | 4 (8)
FATIGUE (ASTHENIA, LETHARGY, MALAISE) (General disorders) | 35 (64)
FEVER (IN THE ABSENCE OF NEUTROPENIA, WHERE NEUTROPENIA IS DEFINED AS ANC <1.0 X 10E9/L) (General disorders) | 9 (13)
FISTULA, PULMONARY/UPPER RESPIRATORY / LUNG (Respiratory, thoracic and mediastinal disorders) | 1 (1)
GASTRITIS (INCLUDING BILE REFLUX GASTRITIS) (Gastrointestinal disorders) | 1 (1)
GASTROINTESTINAL - OTHER (SPECIFY, __) (Gastrointestinal disorders) | 3 (3)
GLUCOSE, SERUM-HIGH (HYPERGLYCEMIA) (Investigations) | 4 (7)
HAIR LOSS/ALOPECIA (SCALP OR BODY) (Skin and subcutaneous tissue disorders) | 14 (14)
HEARING: PATIENTS WITHOUT BASELINE AUDIOGRAM AND NOT ENROLLED IN A MONITORING PROGRAM (Ear and labyrinth disorders) | 1 (1)
HEARTBURN/DYSPEPSIA (Gastrointestinal disorders) | 8 (10)
HEMOGLOBIN (Blood and lymphatic system disorders) | 20 (43)
HEMORRHAGE, GU / BLADDER (Gastrointestinal disorders) | 3 (3)
HEMORRHAGE, PULMONARY/UPPER RESPIRATORY / NOSE (Respiratory, thoracic and mediastinal disorders) | 8 (10)
HEMORRHAGE/BLEEDING - OTHER (SPECIFY, __) (General disorders) | 3 (3)
HEMORRHAGE/BLEEDING ASSOCIATED WITH SURGERY, INTRA-OPERATIVE OR POSTOPERATIVE (Injury, poisoning and procedural complications) | 1 (1)
HICCOUGHS (HICCUPS, SINGULTUS) (Respiratory, thoracic and mediastinal disorders) | 6 (6)
HOT FLASHES/FLUSHES (Endocrine disorders) | 1 (1)
HYPERTENSION (Cardiac disorders) | 14 (19)
HYPOTENSION (Cardiac disorders) | 1 (1)
INFECTION WITH GRADE 3 OR 4 NEUTROPHILS (ANC <1.0 X 10E9/L) / DENTAL-TOOTH (Infections and infestations) | 1 (1)
INFECTION WITH GRADE 3 OR 4 NEUTROPHILS (ANC <1.0 X 10E9/L) / URINARY TRACT NOS (Infections and infestations) | 1 (1)
INFECTION - OTHER (SPECIFY, __) (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / ABDOMEN NOS (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / BLADDER (URINARY) (Infections and infestations) | 2 (3)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / BRONCHUS (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / COLON (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / CONJUNCTIVA (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / EYE NOS (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / RECTUM (Infections and infestations) | 1 (1)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / SINUS (Infections and infestations) | 5 (6)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / SKIN (CELLULITIS) (Infections and infestations) | 2 (2)
INFECTION WITH NORMAL ANC OR GRADE 1 OR 2 NEUTROPHILS / URINARY TRACT NOS (Infections and infestations) | 4 (4)
INFECTION WITH UNKNOWN ANC / SINUS (Infections and infestations) | 1 (1)
INJECTION SITE REACTION/EXTRAVASATION CHANGES (Skin and subcutaneous tissue disorders) | 1 (1)
INSOMNIA (General disorders) | 14 (20)
LEFT VENTRICULAR SYSTOLIC DYSFUNCTION (Cardiac disorders) | 2 (2)
LEUKOCYTES (TOTAL WBC) (Blood and lymphatic system disorders) | 8 (15)
MAGNESIUM, SERUM-LOW (HYPOMAGNESEMIA) (Investigations) | 3 (3)
METABOLIC/LABORATORY - OTHER (SPECIFY, __) (Investigations) | 7 (10)
MOOD ALTERATION / AGITATION (Psychiatric disorders) | 1 (2)
MOOD ALTERATION / ANXIETY (Psychiatric disorders) | 8 (10)
MOOD ALTERATION / DEPRESSION (Psychiatric disorders) | 6 (10)
MUCOSITIS/STOMATITIS (CLINICAL EXAM) / ORAL CAVITY (Surgical and medical procedures) | 9 (10)
MUCOSITIS/STOMATITIS (FUNCTIONAL/SYMPTOMATIC) / ORAL CAVITY (Gastrointestinal disorders) | 4 (5)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / EXTRAOCULAR (Eye disorders) | 1 (1)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / EXTREMITY-UPPER (Musculoskeletal and connective tissue disorders) | 1 (1)
MUSCLE WEAKNESS, GENERALIZED OR SPECIFIC AREA (NOT DUE TO NEUROPATHY) / WHOLE BODY/GENERALIZED (Musculoskeletal and connective tissue disorders) | 4 (4)
MUSCULOSKELETAL/SOFT TISSUE - OTHER (SPECIFY, __) (Musculoskeletal and connective tissue disorders) | 1 (1)
NASAL CAVITY/PARANASAL SINUS REACTIONS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 31 (67)
NEUROLOGY - OTHER (SPECIFY, __) (Nervous system disorders) | 3 (3)
NEUROPATHY: MOTOR (Nervous system disorders) | 2 (3)
NEUROPATHY: SENSORY (Nervous system disorders) | 15 (16)
NEUTROPHILS/GRANULOCYTES (ANC/AGC) (Blood and lymphatic system disorders) | 22 (36)
OCULAR/VISUAL - OTHER (SPECIFY, __) (Eye disorders) | 1 (1)
OPHTHALMOPLEGIA/DIPLOPIA (DOUBLE VISION) (Eye disorders) | 1 (4)
PAIN / ABDOMEN NOS (Gastrointestinal disorders) | 8 (10)
PAIN / ANUS (Gastrointestinal disorders) | 1 (1)
PAIN / BACK (General disorders) | 12 (18)
PAIN / BLADDER (Renal and urinary disorders) | 2 (2)
PAIN / BONE (Musculoskeletal and connective tissue disorders) | 3 (3)
PAIN / CHEST/THORAX NOS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PAIN / DENTAL/TEETH/PERIDONTAL (Gastrointestinal disorders) | 2 (3)
PAIN / EXTERNAL EAR (Ear and labyrinth disorders) | 1 (1)
PAIN / EXTREMITY-LIMB (Musculoskeletal and connective tissue disorders) | 6 (7)
PAIN / HEAD/HEADACHE (General disorders) | 10 (14)
PAIN / JOINT (Musculoskeletal and connective tissue disorders) | 6 (8)
PAIN / KIDNEY (Renal and urinary disorders) | 1 (1)
PAIN / MUSCLE (Musculoskeletal and connective tissue disorders) | 2 (2)
PAIN / PAIN NOS (General disorders) | 1 (1)
PAIN / PELVIS (General disorders) | 2 (2)
PAIN / PENIS (Reproductive system and breast disorders) | 1 (2)
PAIN / PERINEUM (General disorders) | 1 (1)
PAIN / RECTUM (Gastrointestinal disorders) | 1 (2)
PAIN / STOMACH (Gastrointestinal disorders) | 2 (2)
PAIN / THROAT/PHARYNX/LARYNX (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PAIN / URETHRA (Renal and urinary disorders) | 1 (1)
PAIN / VAGINA (Reproductive system and breast disorders) | 1 (4)
PAIN - OTHER (SPECIFY, __) (General disorders) | 10 (15)
PANCREATIC ENDOCRINE: GLUCOSE INTOLERANCE (Endocrine disorders) | 2 (2)
PHLEBITIS (INCLUDING SUPERFICIAL THROMBOSIS) (Vascular disorders) | 2 (2)
PLATELETS (Blood and lymphatic system disorders) | 10 (21)
PNEUMONITIS/PULMONARY INFILTRATES (Respiratory, thoracic and mediastinal disorders) | 1 (1)
POTASSIUM, SERUM-HIGH (HYPERKALEMIA) (Investigations) | 1 (1)
POTASSIUM, SERUM-LOW (HYPOKALEMIA) (Investigations) | 2 (4)
PROTEINURIA (Investigations) | 6 (7)
PRURITUS/ITCHING (Skin and subcutaneous tissue disorders) | 5 (9)
PULMONARY/UPPER RESPIRATORY - OTHER (SPECIFY, __) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
RASH/DESQUAMATION (Skin and subcutaneous tissue disorders) | 2 (2)
RASH: ACNE/ACNEIFORM (Skin and subcutaneous tissue disorders) | 4 (5)
RENAL/GENITOURINARY - OTHER (SPECIFY, __) (Renal and urinary disorders) | 5 (5)
RIGORS/CHILLS (General disorders) | 2 (5)
SODIUM, SERUM-LOW (HYPONATREMIA) (Investigations) | 1 (2)
SWEATING (DIAPHORESIS) (General disorders) | 4 (4)
TASTE ALTERATION (DYSGEUSIA) (Gastrointestinal disorders) | 10 (14)
THROMBOSIS/THROMBUS/EMBOLISM (Vascular disorders) | 4 (5)
THYROID FUNCTION, LOW (HYPOTHYROIDISM) (Endocrine disorders) | 1 (1)
TINNITUS (Ear and labyrinth disorders) | 3 (4)
URINARY FREQUENCY/URGENCY (Renal and urinary disorders) | 5 (5)
URINARY RETENTION (INCLUDING NEUROGENIC BLADDER) (Renal and urinary disorders) | 1 (1)
URINE COLOR CHANGE (Renal and urinary disorders) | 1 (1)
VISION-BLURRED VISION (Eye disorders) | 1 (1)
VISION-PHOTOPHOBIA (Eye disorders) | 1 (1)
VOICE CHANGES/DYSARTHRIA (E.G., HOARSENESS, LOSS OR ALTERATION IN VOICE, LARYNGITIS) (Respiratory, thoracic and mediastinal disorders) | 2 (2)
VOMITING (Gastrointestinal disorders) | 15 (40)
WEIGHT LOSS (General disorders) | 4 (4)
WOUND COMPLICATION, NON-INFECTIOUS (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No